CLINICAL TRIAL: NCT02591186
Title: Effect of Acupuncture on Vascular Biomarkers and Psychological Well-Being of Women Undergoing In Vitro Fertilization (IVF)
Brief Title: Effect of Acupuncture on Vascular Biomarkers and Psychological Well-Being of Women Undergoing IVF
Acronym: AcupunctIVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: L15-117
Record Dates: First submitted 2015-10-07; First posted 2015-10-29 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture arm (Experimental): Participants receiving acupuncture during IVF process
  Interventions: Procedure: Acupuncture
- Control (No Intervention): Control arm not receiving acupuncture during IVF process

INTERVENTIONS:
Procedure: Acupuncture — Participants will receive 3 acupuncture sessions during IVF process
  Arms: Acupuncture arm

SUMMARY:
Experimental Approach: (1) Participants: Women (ages 21 to 42) who seek IVF treatment at the Center for Fertility & Reproductive Surgery will be eligible for the study. Seventy women will be recruited and randomly assigned to either the intervention (acupuncture plus standard care) or the comparison (standard care alone) group. (2) Intervention: Participants in the intervention group will receive 3 acupuncture sessions during the project with the first treatment between day 6-8 of the stimulated IVF cycle, second on the day of embryo transfer and the third one day post transfer. Participants in the comparison group will receive no intervention but will receive standard care. (3) Measures: The primary outcome measures include prostacyclin and thromboxane vasoactive biomarkers. Secondary outcome measures include perceived stress levels. (4) Procedure: Upon IRB approval, an informed consent will be provided to all participants. Pre- and post- acupuncture urinary metabolites of prostacyclin and thromboxane will be assessed. A standardized Perceived Stress Scale will be administered before and after each acupuncture session for the study group, and before and after a 30-40-minute waiting period for the control group.

DETAILED DESCRIPTION:
Hypothesis and Specific Aims

The purpose of this pilot study is to determine if acupuncture affects the vasoactive molecules (prostacyclin and thromboxane) in women undergoing IVF therapy. The investigators' overall hypotheses for this area of study, to be addressed with future research, are: (1) acupuncture augments IVF success by enhancing the perfusion of pelvic organs including the ovaries and the uterus, and (2) acupuncture reduces the levels of stress and optimizes mind-body interaction in individuals undergoing IVF.

Specific Aims:

1. To measure urine prostacyclin and thromboxane, before and after acupuncture, and
2. to assess the impacts of acupuncture on the psychological well-being of women undergoing IVF treatment.

SIGNIFICANCE OF THE STUDY Results from this study will shed light on the mechanism by which acupuncture improves IVF outcomes. This may lead to other treatment strategies to improve success. Likewise, an established mechanism by which acupuncture improves IVF may lead to greater acceptance of this non-conventional treatment modality by the general population.

Research Design and Methods

This is a prospective, randomized, controlled study. Participants will be women in the Principal Investigator's practice seeking IVF. Participants will be randomized 1:1 into either the acupuncture group or the standard of care (no acupuncture) group. Each group will have 3 study visits.

Rationale for the Control Group:

A sham control group is not used because systematic review suggested that sham acupuncture controls may unnecessarily complicate the RCT evidence base given the nature of objective outcomes in IVF study (http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3124624/).

Power analysis

With 35 patients allocated to each group, assuming the Student's T-test will be used to determine the differences between two independent samples, effect sizes d>0.6 will be found statistically significant with alpha .05 and power .80. In practical terms, since the PSS validation samples showed a mean about 13.5 with variance=6.2, only averaged differences greater than 1.5 raw score points in PSS will be found statistically significant.

The investigators plan to seek extramural funding in the future. The investigators will use the data obtained from this pilot study to perform power analysis and to calculate the number of participants needed in future proposals.

ELIGIBILITY:
Inclusion Criteria:

* Women between ages 21-42 years seeking IVF.
* Willing to undergo acupuncture
* No contraindications to needle insertion.

Exclusion Criteria:

* Women currently using alternative therapies such as acupressure, herbal supplements and meditation techniques.
* Women with generalized psoriasis, neuropathy or coagulopathies posing increased risk due to needle insertion.
* Women with previous experience with acupuncture.

***Please note that we are unable to give a discount on IVF cost for participating in the study.***

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Urine prostacyclin before and after acupuncture | Within 8-week course of IVF treatment
  Measurement of the vasoactive molecule prostacyclin (pg/mg creatinine) in women undergoing IVF therapy.
Urine thromboxane before and after acupuncture | Within 8-week course of IVF treatment
  Measurement of the vasoactive molecule thromboxane (pg/mg creatinine) in women undergoing IVF therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Phy, DO, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech Health Science Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Lim H, Paria BC, Das SK, Dinchuk JE, Langenbach R, Trzaskos JM, Dey SK. Multiple female reproductive failures in cyclooxygenase 2-deficient mice. Cell. 1997 Oct 17;91(2):197-208. doi: 10.1016/s0092-8674(00)80402-x. PMID 9346237
- [Background] Pandian Z, Bhattacharya S, Ozturk O, Serour G, Templeton A. Number of embryos for transfer following in-vitro fertilisation or intra-cytoplasmic sperm injection. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003416. doi: 10.1002/14651858.CD003416.pub3. PMID 19370588
- [Background] Anderson BJ, Haimovici F, Ginsburg ES, Schust DJ, Wayne PM. In vitro fertilization and acupuncture: clinical efficacy and mechanistic basis. Altern Ther Health Med. 2007 May-Jun;13(3):38-48. PMID 17515023
- [Background] Manheimer E, Zhang G, Udoff L, Haramati A, Langenberg P, Berman BM, Bouter LM. Effects of acupuncture on rates of pregnancy and live birth among women undergoing in vitro fertilisation: systematic review and meta-analysis. BMJ. 2008 Mar 8;336(7643):545-9. doi: 10.1136/bmj.39471.430451.BE. Epub 2008 Feb 7. PMID 18258932
- [Background] Huang JC, Wun WS, Goldsby JS, Egan K, FitzGerald GA, Wu KK. Prostacyclin receptor signaling and early embryo development in the mouse. Hum Reprod. 2007 Nov;22(11):2851-6. doi: 10.1093/humrep/dem304. Epub 2007 Sep 28. PMID 17905746
- [Background] Huang JC, Goldsby JS, Wun WS. Prostacyclin enhances the implantation and live birth potentials of mouse embryos. Hum Reprod. 2004 Aug;19(8):1856-60. doi: 10.1093/humrep/deh352. Epub 2004 Jun 17. PMID 15205402
- [Background] Ruan KH, Deng H, So SP. Engineering of a protein with cyclooxygenase and prostacyclin synthase activities that converts arachidonic acid to prostacyclin. Biochemistry. 2006 Nov 28;45(47):14003-11. doi: 10.1021/bi0614277. PMID 17115695
- [Background] Majerus PW. Arachidonate metabolism in vascular disorders. J Clin Invest. 1983 Nov;72(5):1521-5. doi: 10.1172/JCI111110. No abstract available. PMID 6313764
- [Background] Samuelsson B, Goldyne M, Granstrom E, Hamberg M, Hammarstrom S, Malmsten C. Prostaglandins and thromboxanes. Annu Rev Biochem. 1978;47:997-1029. doi: 10.1146/annurev.bi.47.070178.005025. No abstract available. PMID 209733
- [Background] Smith WL. Prostaglandin biosynthesis and its compartmentation in vascular smooth muscle and endothelial cells. Annu Rev Physiol. 1986;48:251-62. doi: 10.1146/annurev.ph.48.030186.001343. PMID 3085582
- [Background] Funk CD. Prostaglandins and leukotrienes: advances in eicosanoid biology. Science. 2001 Nov 30;294(5548):1871-5. doi: 10.1126/science.294.5548.1871. PMID 11729303
- [Background] Ruan KH. Advance in understanding the biosynthesis of prostacyclin and thromboxane A2 in the endoplasmic reticulum membrane via the cyclooxygenase pathway. Mini Rev Med Chem. 2004 Aug;4(6):639-47. doi: 10.2174/1389557043403710. PMID 15279598
- [Background] Ruan KH, Dogne JM. Implications of the molecular basis of prostacyclin biosynthesis and signaling in pharmaceutical designs. Curr Pharm Des. 2006;12(8):925-41. doi: 10.2174/138161206776055994. PMID 16533160
- [Background] Dogne JM, Hanson J, de Leval X, Pratico D, Pace-Asciak CR, Drion P, Pirotte B, Ruan KH. From the design to the clinical application of thromboxane modulators. Curr Pharm Des. 2006;12(8):903-23. doi: 10.2174/138161206776055921. PMID 16533159
- [Background] Needleman P, Turk J, Jakschik BA, Morrison AR, Lefkowith JB. Arachidonic acid metabolism. Annu Rev Biochem. 1986;55:69-102. doi: 10.1146/annurev.bi.55.070186.000441. No abstract available. PMID 3017195
- [Background] Bunting S, Gryglewski R, Moncada S, Vane JR. Arterial walls generate from prostaglandin endoperoxides a substance (prostaglandin X) which relaxes strips of mesenteric and coeliac ateries and inhibits platelet aggregation. Prostaglandins. 1976 Dec;12(6):897-913. doi: 10.1016/0090-6980(76)90125-8. PMID 1005741
- [Background] Moncada S, Herman AG, Higgs EA, Vane JR. Differential formation of prostacyclin (PGX or PGI2) by layers of the arterial wall. An explanation for the anti-thrombotic properties of vascular endothelium. Thromb Res. 1977 Sep;11(3):323-44. doi: 10.1016/0049-3848(77)90185-2. No abstract available. PMID 335560
- [Background] Weksler BB, Ley CW, Jaffe EA. Stimulation of endothelial cell prostacyclin production by thrombin, trypsin, and the ionophore A 23187. J Clin Invest. 1978 Nov;62(5):923-30. doi: 10.1172/JCI109220. PMID 361756
- [Background] Ingerman-Wojenski C, Silver MJ, Smith JB, Macarak E. Bovine endothelial cells in culture produce thromboxane as well as prostacyclin. J Clin Invest. 1981 May;67(5):1292-6. doi: 10.1172/jci110157. PMID 7014633
- [Background] Smith WL, DeWitt DL, Allen ML. Bimodal distribution of the prostaglandin I2 synthase antigen in smooth muscle cells. J Biol Chem. 1983 May 10;258(9):5922-6. PMID 6406508
- [Background] Coceani F, Ackerley C, Seidlitz E, Kelsey L. Function of cyclo-oxygenase-1 and cyclo-oxygenase-2 in the ductus arteriosus from foetal lamb: differential development and change by oxygen and endotoxin. Br J Pharmacol. 2001 Jan;132(1):241-51. doi: 10.1038/sj.bjp.0703779. PMID 11156583
- [Background] Pakrasi PL, Jain AK. Cyclooxygenase-2-derived endogenous prostacyclin reduces apoptosis and enhances embryo viability in mouse. Prostaglandins Leukot Essent Fatty Acids. 2008 Jul-Aug;79(1-2):27-33. doi: 10.1016/j.plefa.2008.07.006. Epub 2008 Sep 3. PMID 18771909
- [Background] Stener-Victorin E, Waldenstrom U, Andersson SA, Wikland M. Reduction of blood flow impedance in the uterine arteries of infertile women with electro-acupuncture. Hum Reprod. 1996 Jun;11(6):1314-7. doi: 10.1093/oxfordjournals.humrep.a019378. PMID 8671446
- [Background] Uchida S, Hotta H. Acupuncture affects regional blood flow in various organs. Evid Based Complement Alternat Med. 2008 Jun;5(2):145-51. doi: 10.1093/ecam/nem051. PMID 18604254
- [Background] Zhang S, Ye X, Shan Q, Zhang W, Ye L, Cui Y. Effects of acupuncture on the levels of endothelin, TXB2, and 6-keto-PGF1 alpha in apoplexy patients. J Tradit Chin Med. 1999 Mar;19(1):39-43. PMID 10453582
- [Background] Xu N. [Effect of electroacupuncture at "taixi" point on plasma thromboxane A2 and prostacyclin in the rabbit with renal ischemia]. Zhen Ci Yan Jiu. 1993;18(3):240-2. Chinese. PMID 7923725
- [Background] Yuan J, Westney OL, Ruan KH, Wang R. A new strategy, SuperEnzyme gene therapy in penile rehabilitation. J Sex Med. 2009 Mar;6 Suppl 3:328-33. doi: 10.1111/j.1743-6109.2008.01191.x. PMID 19267856
- [Background] Ruan KH, So SP, Cervantes V, Wu H, Wijaya C, Jentzen RR. An active triple-catalytic hybrid enzyme engineered by linking cyclo-oxygenase isoform-1 to prostacyclin synthase that can constantly biosynthesize prostacyclin, the vascular protector. FEBS J. 2008 Dec;275(23):5820-9. doi: 10.1111/j.1742-4658.2008.06703.x. PMID 19021758
- [Background] Ruan KH, So SP, Wu H, Cervantes V. Large-scale expression, purification, and characterization of an engineered prostacyclin-synthesizing enzyme with therapeutic potential. Arch Biochem Biophys. 2008 Dec 1;480(1):41-50. doi: 10.1016/j.abb.2008.09.010. Epub 2008 Sep 22. PMID 18835243
- [Background] Ruan KH, Wu J, Cervantes V. Characterization of the substrate mimic bound to engineered prostacyclin synthase in solution using high-resolution NMR spectroscopy and mutagenesis: implication of the molecular mechanism in biosynthesis of prostacyclin. Biochemistry. 2008 Jan 15;47(2):680-8. doi: 10.1021/bi701671q. Epub 2007 Dec 15. PMID 18081314
- [Background] Ruan KH, Deng H, Wu J, So SP. The N-terminal membrane anchor domain of the membrane-bound prostacyclin synthase involved in the substrate presentation of the coupling reaction with cyclooxygenase. Arch Biochem Biophys. 2005 Mar 15;435(2):372-81. doi: 10.1016/j.abb.2004.12.018. PMID 15708381
- [Background] Ni F, So SP, Cervantes V, Ruan KH. A profile of the residues in the second extracellular loop that are critical for ligand recognition of human prostacyclin receptor. FEBS J. 2008 Jan;275(1):128-37. doi: 10.1111/j.1742-4658.2007.06183.x. Epub 2007 Nov 27. PMID 18042246
- [Background] Zhang L, Bastepe M, Juppner H, Ruan KH. Characterization of the molecular mechanisms of the coupling between intracellular loops of prostacyclin receptor with the C-terminal domain of the Galphas protein in human coronary artery smooth muscle cells. Arch Biochem Biophys. 2006 Oct 1;454(1):80-8. doi: 10.1016/j.abb.2006.06.023. Epub 2006 Jul 25. PMID 16942748
- [Background] Zhang L, Wu J, Ruan KH. Solution structure of the first intracellular loop of prostacyclin receptor and implication of its interaction with the C-terminal segment of G alpha s protein. Biochemistry. 2006 Feb 14;45(6):1734-44. doi: 10.1021/bi0515669. PMID 16460020
- [Background] Ruan CH, Wu J, Ruan KH. A strategy using NMR peptide structures of thromboxane A2 receptor as templates to construct ligand-recognition pocket of prostacyclin receptor. BMC Biochem. 2005 Nov 4;6:23. doi: 10.1186/1471-2091-6-23. PMID 16271145
- [Background] Zhang L, Huang G, Wu J, Ruan KH. A profile of the residues in the first intracellular loop critical for Gs-mediated signaling of human prostacyclin receptor characterized by an integrative approach of NMR-experiment and mutagenesis. Biochemistry. 2005 Aug 30;44(34):11389-401. doi: 10.1021/bi050483p. PMID 16114876
- [Background] Ruan KH, Wu J, So SP, Jenkins LA. Evidence of the residues involved in ligand recognition in the second extracellular loop of the prostacyclin receptor characterized by high resolution 2D NMR techniques. Arch Biochem Biophys. 2003 Oct 1;418(1):25-33. doi: 10.1016/s0003-9861(03)00401-6. PMID 13679079
- [Background] Ruan KH, Wu J, Wang LH. Solution structure of a common substrate mimetic of cyclooxygenase-downstream synthases bound to an engineered thromboxane A2 synthase using a high-resolution NMR technique. Arch Biochem Biophys. 2005 Dec 15;444(2):165-73. doi: 10.1016/j.abb.2005.10.010. Epub 2005 Nov 2. PMID 16297851
- [Background] So SP, Li D, Ruan KH. Identification of the substrate interaction site in the N-terminal membrane anchor segment of thromboxane A2 synthase by determination of its substrate analog conformational changes using high resolution NMR technique. J Biol Chem. 2000 Dec 29;275(52):40679-85. doi: 10.1074/jbc.M005752200. PMID 11006279
- [Background] Ruan KH, Li D, Ji J, Lin YZ, Gao X. Structural characterization and topology of the second potential membrane anchor region in the thromboxane A2 synthase amino-terminal domain. Biochemistry. 1998 Jan 20;37(3):822-30. doi: 10.1021/bi971881y. PMID 9454571
- [Background] Ruan KH, Cervantes V, Wu J. Ligand-specific conformation determines agonist activation and antagonist blockade in purified human thromboxane A2 receptor. Biochemistry. 2009 Apr 14;48(14):3157-65. doi: 10.1021/bi801443g. PMID 19170518
- [Background] Ruan KH, Wijaya C, Cervantes V, Wu J. Characterization of the prostaglandin H2 mimic: binding to the purified human thromboxane A2 receptor in solution. Arch Biochem Biophys. 2008 Sep 15;477(2):396-403. doi: 10.1016/j.abb.2008.05.022. Epub 2008 Jun 17. PMID 18590695
- [Background] Ruan KH, Cervantes V, Wu J. A simple, quick, and high-yield preparation of the human thromboxane A2 receptor in full size for structural studies. Biochemistry. 2008 Jul 1;47(26):6819-26. doi: 10.1021/bi702501g. Epub 2008 Jun 5. PMID 18529068
- [Background] Wu J, Feng M, Ruan KH. Assembling NMR structures for the intracellular loops of the human thromboxane A2 receptor: implication of the G protein-coupling pocket. Arch Biochem Biophys. 2008 Feb 1;470(1):73-82. doi: 10.1016/j.abb.2007.11.016. Epub 2007 Dec 3. PMID 18073117
- [Background] Ruan KH, Wu J, So SP, Jenkins LA, Ruan CH. NMR structure of the thromboxane A2 receptor ligand recognition pocket. Eur J Biochem. 2004 Jul;271(14):3006-16. doi: 10.1111/j.1432-1033.2004.04232.x. PMID 15233797
- [Background] Geng L, Wu J, So SP, Huang G, Ruan KH. Structural and functional characterization of the first intracellular loop of human thromboxane A2 receptor. Arch Biochem Biophys. 2004 Mar 15;423(2):253-65. doi: 10.1016/j.abb.2004.01.001. PMID 15001390
- [Background] Wu J, So SP, Ruan KH. Solution structure of the third extracellular loop of human thromboxane A2 receptor. Arch Biochem Biophys. 2003 Jun 15;414(2):287-93. doi: 10.1016/s0003-9861(03)00192-9. PMID 12781781
- [Background] So SP, Wu J, Huang G, Huang A, Li D, Ruan KH. Identification of residues important for ligand binding of thromboxane A2 receptor in the second extracellular loop using the NMR experiment-guided mutagenesis approach. J Biol Chem. 2003 Mar 28;278(13):10922-7. doi: 10.1074/jbc.M209337200. Epub 2003 Jan 27. PMID 12551898
- [Background] Ruan KH, Cervantes V, So SP. Engineering of a novel hybrid enzyme: an anti-inflammatory drug target with triple catalytic activities directly converting arachidonic acid into the inflammatory prostaglandin E2. Protein Eng Des Sel. 2009 Dec;22(12):733-40. doi: 10.1093/protein/gzp058. Epub 2009 Oct 22. PMID 19850676
- [Background] Chillar A, Wu J, So SP, Ruan KH. Involvement of non-conserved residues important for PGE2 binding to the constrained EP3 eLP2 using NMR and site-directed mutagenesis. FEBS Lett. 2008 Aug 20;582(19):2863-8. doi: 10.1016/j.febslet.2008.07.018. Epub 2008 Jul 22. PMID 18652829
- [Background] Huang JC, Arbab F, Tumbusch KJ, Goldsby JS, Matijevic-Aleksic N, Wu KK. Human fallopian tubes express prostacyclin (PGI) synthase and cyclooxygenases and synthesize abundant PGI. J Clin Endocrinol Metab. 2002 Sep;87(9):4361-8. doi: 10.1210/jc.2002-020199. PMID 12213900
- [Background] Arbab F, Goldsby J, Matijevic-Aleksic N, Huang G, Ruan KH, Huang JC. Prostacyclin is an autocrine regulator in the contraction of oviductal smooth muscle. Hum Reprod. 2002 Dec;17(12):3053-9. doi: 10.1093/humrep/17.12.3053. PMID 12456602
- [Background] Huang JC, Goldsby JS, Arbab F, Melhem Z, Aleksic N, Wu KK. Oviduct prostacyclin functions as a paracrine factor to augment the development of embryos. Hum Reprod. 2004 Dec;19(12):2907-12. doi: 10.1093/humrep/deh520. Epub 2004 Oct 18. PMID 15492023
- [Background] Huang JC, Wun WS, Goldsby JS, Matijevic-Aleksic N, Wu KK. Cyclooxygenase-2-derived endogenous prostacyclin enhances mouse embryo hatching. Hum Reprod. 2004 Dec;19(12):2900-6. doi: 10.1093/humrep/deh524. Epub 2004 Oct 15. PMID 15489241
- [Background] Huang JC, Wun WS, Goldsby JS, Wun IC, Noorhasan D, Wu KK. Stimulation of embryo hatching and implantation by prostacyclin and peroxisome proliferator-activated receptor delta activation: implication in IVF. Hum Reprod. 2007 Mar;22(3):807-14. doi: 10.1093/humrep/del429. Epub 2006 Nov 17. PMID 17114194
- [Background] de Lacey S, Smith CA, Paterson C. Building resilience: a preliminary exploration of women's perceptions of the use of acupuncture as an adjunct to In Vitro Fertilisation. BMC Complement Altern Med. 2009 Dec 12;9:50. doi: 10.1186/1472-6882-9-50. PMID 20003370
- [Background] Ng EH, So WS, Gao J, Wong YY, Ho PC. The role of acupuncture in the management of subfertility. Fertil Steril. 2008 Jul;90(1):1-13. doi: 10.1016/j.fertnstert.2008.02.094. Epub 2008 Apr 28. PMID 18440533
- [Background] Stener-Victorin E, Humaidan P. Use of acupuncture in female infertility and a summary of recent acupuncture studies related to embryo transfer. Acupunct Med. 2006 Dec;24(4):157-63. doi: 10.1136/aim.24.4.157. PMID 17264833
- [Background] Ho M, Huang LC, Chang YY, Chen HY, Chang WC, Yang TC, Tsai HD. Electroacupuncture reduces uterine artery blood flow impedance in infertile women. Taiwan J Obstet Gynecol. 2009 Jun;48(2):148-51. doi: 10.1016/S1028-4559(09)60276-X. PMID 19574177
- [Background] Huang JC, Wun WS, Goldsby JS, Wun IC, Falconi SM, Wu KK. Prostacyclin enhances embryo hatching but not sperm motility. Hum Reprod. 2003 Dec;18(12):2582-9. doi: 10.1093/humrep/deg490. PMID 14645174
- [Background] Urbich C, Kuehbacher A, Dimmeler S. Role of microRNAs in vascular diseases, inflammation, and angiogenesis. Cardiovasc Res. 2008 Sep 1;79(4):581-8. doi: 10.1093/cvr/cvn156. Epub 2008 Jun 11. PMID 18550634
- [Background] Planat-Benard V, Silvestre JS, Cousin B, Andre M, Nibbelink M, Tamarat R, Clergue M, Manneville C, Saillan-Barreau C, Duriez M, Tedgui A, Levy B, Penicaud L, Casteilla L. Plasticity of human adipose lineage cells toward endothelial cells: physiological and therapeutic perspectives. Circulation. 2004 Feb 10;109(5):656-63. doi: 10.1161/01.CIR.0000114522.38265.61. Epub 2004 Jan 20. PMID 14734516
- [Derived] Zhang Y, Phy J, Scott-Johnson C, Garos S, Orlando J, Prien S, Huang JC. Effects of a Delphi consensus acupuncture treatment protocol on the levels of stress and vascular tone in women undergoing in-vitro fertilization: a randomized clinical trial protocol. BMC Complement Altern Med. 2017 Apr 4;17(1):197. doi: 10.1186/s12906-017-1693-4. PMID 28376836

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT02591186/Prot_SAP_000.pdf